CLINICAL TRIAL: NCT05159908
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled, Dose-Finding Study to Investigate Safety, Tolerability, Pharmacokinetics, and Efficacy of NBI-921352 as Adjunctive Therapy in Adult Subjects With Focal Onset Seizures (FOS)
Brief Title: A Study to Investigate How Effective, Safe and Tolerable the Drug NBI-921352 is When Used With Anti-seizure Medications in Adults With Focal Onset Seizures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NBI-921352-FOS2021; 2021-001433-39 (EudraCT Number)
Record Dates: First submitted 2021-11-30; First posted 2021-12-16 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Focal Onset Seizure; Focal Onset Epilepsy
Keywords: Epilepsy; focal seizure; sodium channel; voltage-gated; alpha subunit; Nav1.6 inhibitor; Antiseizure medication; ASM; Antiepileptic drug; AED; partial seizure; partial onset epilepsy
MeSH Terms: conditions — Seizures; Epilepsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo schedule (Placebo Comparator): Participant follows Placebo schedule (13 weeks)
  Interventions: Drug: Placebo
- Dose schedule A (Experimental): Participant follows Dose schedule A (13 weeks)
  Interventions: Drug: NBI-921352
- Dose schedule B (Experimental): Participant follows Dose schedule B (13 weeks)
  Interventions: Drug: NBI-921352
- Dose schedule C (Experimental): Participant follows Dose schedule C (13 weeks)
  Interventions: Drug: NBI-921352

INTERVENTIONS:
Drug: NBI-921352 — Tablets for oral administration
  Arms: Dose schedule A; Dose schedule B; Dose schedule C
Drug: Placebo — Matching placebo tablets for oral administration
  Arms: Placebo schedule

SUMMARY:
This study will evaluate the safety, pharmacokinetics, and efficacy of three different doses of NBI-921352 versus placebo in adults with focal onset seizures

ELIGIBILITY:
Key Inclusion Criteria:

1. Capable of providing consent and has completed the written informed consent.
2. Male or female, 18 to 65 years of age, inclusive, with a body mass index (BMI) < 40 kg/m^2.
3. Diagnosis of focal onset epilepsy according to the International League Against Epilepsy (ILAE) Classification of Epilepsy (2017) at least 18 months before screening.
4. History of uncontrolled seizures despite adequate treatment with at least 1 anti-seizure medication (ASM) for at least 18 months prior to screening.
5. Treatment with at least 1 but not more than 4 ASMs for at least 1 month before screening, during the baseline seizure diary data collection, and throughout the duration of the study.
6. Be able to keep accurate seizure diaries.
7. Documented seizure frequency in the baseline seizure diary of ≥8 countable focal seizures during the 8-week seizure baseline period.

Key Exclusion Criteria:

1. History of epilepsy with only nonmotor seizures without an observable component, psychogenic nonepileptic seizures, or primary generalized seizures.
2. Presence or previous history of developmental and/or epileptic encephalopathy.
3. Presence of seizure types other than FOS.
4. Status epilepticus within the last 12 months before enrollment.
5. Any suicidal behavior or suicidal ideation of type 4 (active suicidal ideation with some intent to act, without specific plan) or type 5 (active suicidal ideation with specific plan and intent) based on the C-SSRS in the 2 years before screening, a history of suicide attempt in the last 2 years, or more than 1 lifetime suicide attempt.
6. Multiple drug allergies or a severe drug reaction to an ASM(s), including dermatological (eg, Stevens-Johnson syndrome), hematological, or organ toxicity reactions.
7. An implanted responsive neurostimulator system (RNS).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2023-08-21 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Serious Treatment-emergent Adverse Events (TEAEs), TEAEs Leading to Discontinuation of Study Treatment, and Fatal TEAEs | Through Week 15
NBI-921352 exposure-efficacy response relationship, defined as the slope of the relationship between reduction in monthly focal onset seizure frequency and plasma concentration at steady state | Baseline to Week 11

SECONDARY OUTCOMES:
Percent Change from Baseline in Monthly Focal Onset Seizure Frequency During the Treatment Period | Baseline and Weeks 1 to 11
Percent Change from Baseline in Monthly Focal Onset Seizure Frequency During the Maintenance period | Baseline and Weeks 4 to 11
Clinical Global Impression of Change (CGIC) Scores at Week 11 | Week 11
Percentage of Participants with a ≥ 50% reduction in monthly (28 days) focal onset seizure frequency during the treatment period | Baseline and Weeks 1 to 11

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Lead, Study Director — Neurocrine Biosciences
Locations (25):
- Australia (5):
  - Neurocrine Clinical Site, Randwick, New South Wales
  - Neurocrine Clinical Site, Ivanhoe, Victoria
  - Neurocrine Clinical Site, Melbourne, Victoria
  - Neurocrine Clinical Site, Parkville, Victoria
  - Neurocrine Clinical Site, Prahran, Victoria
- Belgium (3):
  - Neurocrine Clinical Site, Brussels
  - Neurocrine Clinical Site, Ghent
  - Neurocrine Clinical Site, Leuven
- Czechia (4):
  - Neurocrine Clinical Site, Brno
  - Neurocrine Clinical Site, Ostrava
  - Neurocrine Clinical Site, Prague
  - Neurocrine Clinical Site, Rychnov nad Kněžnou
- France (4):
  - Neurocrine Clinical Site, Bron
  - Neurocrine Clinical Site, Lille
  - Neurocrine Clinical Site, Rennes
  - Neurocrine Clinical Site, Toulouse
- Hungary (3):
  - Neurocrine Clinical Site, Budapest
  - Neurocrine Clinical Site, Debrecen
  - Neurocrine Clinical Site, Pécs
- Italy (3):
  - Neurocrine Clinical Site, Bologna
  - Neurocrine Clinical Site, Milan
  - Neurocrine Clinical Site, Pavia
- Spain (3):
  - Neurocrine Clinical Site, Barcelona
  - Neurocrine Clinical Site, Madrid
  - Neurocrine Clinical Site, Valencia

IPD SHARING:
Plan to Share IPD: No